CLINICAL TRIAL: NCT00671749
Title: A Clinical Assessment of Combination Therapy With Differin® Gel, 0.3% With Duac® (Clindamycin/Benzoyl Peroxide Gel) in Subjects With Acne Vulgaris
Brief Title: Combination Therapy With Differin® Gel 0.3% and Duac® (Clindamycin/Benzoyl Peroxide Gel) in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US10066
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2016-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Treatment (Experimental): adapalene gel, 0.3%
  Other Names:
  Differin® Gel, 0.3% Applied once daily at bedtime
  clindamycin/benzoyl peroxide gel
  Other Names:
  Duac® Gel Applied once daily in the morning
  Interventions: Drug: adapalene gel, 0.3%; Drug: clindamycin/benzoyl peroxide gel

INTERVENTIONS:
Drug: adapalene gel, 0.3% — Applied once daily at bedtime
  Other Names: Differin® Gel, 0.3%
Drug: clindamycin/benzoyl peroxide gel — Applied once daily in the morning
  Other Names: Duac® Gel

SUMMARY:
This study is to determine the efficacy and safety of 12 week treatment with Differin® Gel 0.3% applied in the evening, in combination with Duac® (Clindamycin/Benzoyl Peroxide Gel) applied in the morning, in Subjects with Acne vulgaris.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a minimum of 20 inflammatory lesions on the face;
2. Subjects with a minimum of 15 and a maximum of 100 non-inflammatory lesions (open and closed comedones) on the face, excluding the nose;
3. Subject has a Global Severity Assessment

Exclusion Criteria:

1. Subjects with more than three nodulo-cystic lesions

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron W Gottschalk, MD, Study Director — Galderma R&D
Locations (4):
- United States (4):
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Derm Research, P.L.L.C., Louisville, Kentucky
  - Brodell Medical, Warren, Ohio
  - Northwest Cutaneous Research Specialists, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Therapy: Each subject applied each of the study medications once daily: Duac® Topical Gel in the morning and Differin® Gel, 0.3% in the evening.
Period: Overall Study
Arm/Group | Combination Therapy
Started | 100
Completed | 92
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.2 (5.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 77
  More than one race | 10
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 0
Duration of Acne [Mean (Standard Deviation); unit: years] | 4.0 (3.91)
Fitzpatrick Skin Type [Number; unit: participants] — Investigator assessment based on the standard Fitzpatrick Skin Test (Scale I to VI). Example:
  TYPE 1: Highly sensitive, always burns, never tans. TYPE 2: Very sun sensitive, burns easily, tans minimally. TYPE 3: Sun sensitive skin, sometimes burns, slowly tans to light brown. TYPE 4: Minimally sun sensitive, burns minimally, always tans to moderate brown.
  TYPE 5: Sun insensitive skin, rarely burns, tans well. TYPE 6: Sun insensitive, never burns, deeply pigmented
  participants
    I | 1
    II | 27
    III | 38
    IV | 22
    V | 4
    VI | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Lesion Counts
Time Frame: 6 and 12 weeks
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy
Number analyzed (Participants) | 100
Percent Change
  Week 6 | -47 (24.43)
  Week 12 | -64 (24.07)

2. Secondary Outcome: Global Severity Assessment Success
Description: Global Severity was assessed on a 6 point scale (Clear, Almost Clear, Mild, Moderate, Severe). The scale was dichotomized to success or failure where success = Clear or Almost Clear
Time Frame: 6 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 100
participants
  Week 6 | 8
  Week 12 | 42

3. Secondary Outcome: Global Assessment of Improvement From Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 100
participants
  Clear | 3
  Almost Clear | 40
  Marked Improvement | 27
  Moderate Improvement | 16
  Minimal Improvement | 5
  No Change | 8
  Worse | 1

4. Secondary Outcome: Worst Post Baseline Tolerability Assessment - Erythema
Description: Please Note: "Tolerability Assessments" were captured separately from adverse events. Tolerability changes that required a dose modification or concomitant treatment were to be recorded on the Adverse Event CRF.
Time Frame: 12 weeks
Population: Safety Population (n=99)
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 99
participants
  None | 29
  Mild | 37
  Moderate | 33
  Severe | 0

5. Secondary Outcome: Worst Post Baseline Tolerability Assessment - Scaling
Description: as for outcome 4
Time Frame: 12 weeks
Population: Safety Population (n=99)
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 99
participants
  None | 53
  Mild | 27
  Moderate | 16
  Severe | 3

6. Secondary Outcome: Worst Post Baseline Tolerability Assessment - Dryness
Description: as for outcome 4
Time Frame: 12 weeks
Population: Safety Population (n=99)
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 99
participants
  None | 49
  Mild | 27
  Moderate | 20
  Severe | 3

7. Secondary Outcome: Worst Post Baseline Tolerability Assessment - Burning/Stinging
Description: as for outcome 4
Time Frame: 12 weeks
Population: Safety Population (n=99)
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 99
participants
  None | 67
  Mild | 18
  Moderate | 9
  Severe | 5

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Please Note: "Tolerability Assessments" were captured separately from adverse events. Tolerability changes that required a dose modification or concomitant treatment were to be recorded on the Adverse Event CRF.
Arm/Group | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 32/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=99)
Application Site Burn (General disorders) | 32
Application Site Dryness (General disorders) | 24
Application Site Erythema (General disorders) | 10
Application Site Exfoliation (General disorders) | 7
Application Site Discomfort (General disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days